CLINICAL TRIAL: NCT06117371
Title: A Two-phase, Multicenter, Open Phase I Study of BEBT-607 Tablets in The Treatment of Advanced or Metastatic Solid Tumors With KRAS G12C Mutation
Brief Title: Study of BEBT-607 Tablets in The Treatment of Advanced or Metastatic Solid Tumors With KRAS G12C Mutation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeBetter Med Inc (Industry)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-607-P01
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Advanced or Metastatic Solid Tumor; KRAS G12C Mutation
Keywords: BEBT-607; Safety; Tolerance; effectiveness; Pharmacokinetics
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Phase Ⅰa:
  Six dose levels are carried out, and the initial dose of BEBT-607 tablets is set as 100mg/ day. The climbing study is carried out by accelerated titration method combined with "3+3" mode.
  Phase Ⅰb:
  According to the pharmacokinetics, safety, and preliminary efficacy results of phase Ⅰa , one to three cohorts with target dose or tumor species are selected for dose extension trial, in which participants receive continuous administration of the experimental drug BEBT-607 tablets until disease progression or toxicity became intolerable or patients stopped or died.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Monotherapy group 1 (Experimental): BEBT-607 tablets, 100mg/day,50mg each time, are administered once a day in the single administration phase and twice a day in the continuous administration phase (only once on the 28th day of the first cycle) for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 2 (Experimental): BEBT-607 tablets, 200mg/day,100mg each time, are administered once a day in the single administration phase and twice a day in the continuous administration phase (only once on the 28th day of the first cycle) for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 3 (Experimental): BEBT-607 tablets, 300mg/day,150mg each time, are administered once a day in the single administration phase and twice a day in the continuous administration phase (only once on the 28th day of the first cycle) for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 4 (Experimental): BEBT-607 tablets, 400mg/day,200mg each time, are administered once a day in the single administration phase and twice a day in the continuous administration phase (only once on the 28th day of the first cycle) for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 5 (Experimental): BEBT-607 tablets, 600mg/day,300mg each time, are administered once a day in the single administration phase and twice a day in the continuous administration phase (only once on the 28th day of the first cycle) for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 6 (Experimental): BEBT-607 tablets, 800mg/day,400mg each time, are administered once a day in the single administration phase and twice a day in the continuous administration phase (only once on the 28th day of the first cycle) for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 7 (Experimental): BEBT-607 tablets, 300mg/day,150mg each time, are administered twice a day (only once on day 1 and day 28 of the first cycle), continuous administration for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 8 (Experimental): BEBT-607 tablets, 400mg/day,200mg each time, are administered twice a day (only once on day 1 and day 28 of the first cycle), continuous administration for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets
- Monotherapy group 9 (Experimental): BEBT-607 tablets, 600mg/day,300mg each time, are administered twice a day (only once on day 1 and day 28 of the first cycle), continuous administration for 28 days. 28 days is as a treatment cycle.
  Interventions: Drug: BEBT-607Tablets

INTERVENTIONS:
Drug: BEBT-607Tablets — PhaseⅠa:100mg,200mg,300mg,400mg,600mg or 800mg/day,50mg,100mg,150mg,200mg,300mg or 400mg each time, once a day in the single administration phase and twice a day in the continuous administration phase (only once on the 28th day of the first cycle) for 28 days,28 days is as a treatment cycle.
  PhaseⅠb:300mg,400mg or 600mg/day, 150mg,200mg or 300mg each time,twice a day (only once on day 1 and day 28 of the first cycle), continuous administration for 28 days,28 days is as a treatment cycle.
  Other Names: C200825009-FP

SUMMARY:
This is a two-phase, multicenter, open phase I clinical study, with phase Ia as dose escalation phase and phase Ib as dose expansion phase, to evaluate the safety tolerability and pharmacokinetic characteristics of BEBT-607 tablets in patients with advanced or metastatic solid tumors associated with KRAS G12C mutation. To evaluate the efficacy of BEBT-607 tablets in the treatment of patients with advanced or metastatic solid tumors with KRAS G12C mutation, and to determine the recommended dose (RP2D) for Phase II clinical trials of BEBT-607 tablets in patients with advanced or metastatic solid tumors with KRAS G12C mutation.

DETAILED DESCRIPTION:
Phase Ⅰa:

The dose escalation plan is to carry out about 6 dose levels. The initial dose of BEBT-607 tablets is set at 100mg/ day, and the subsequent dose groups are first increased by 100%. If a case of drug-related grade 2 non-hematological toxicity or grade 3 hematological toxicity is found and does not reach DLT, the subsequent dose groups are increased by 50%. If one case of dose limiting toxicity(DLT) is found and does not reach maximum tolerated dose(MTD ), the subsequent dose group is increased by 33%（Doses are rounded to multiples of 100mg）.The single dose is 1/2 of the total daily dose, and the single administration phase is administered once a day, and the continuous administration phase is administered twice a day (only once on the 28th day of the first cycle).

Phase Ⅰb:

According to the pharmacokinetics, safety and preliminary efficacy results of phase Ⅰa dose escalation phase, one to three cohorts with target dose or tumor species are selected for dose extension trial, and a maximum of 30 subjects are enrolled in each cohort. The subjects receive BEBT-607 tablets twice a day, orally before breakfast and before dinner, respectively. There is a treatment cycle every 28 days (On days 1 and 28 of the first cycle, the drug is administered only once before breakfast). The study process for each subject consisted of three phases: screening, treatment, and follow-up. During treatment, participants are required to undergo safety checks every four weeks from the first dose, tumor assessments every eight weeks, safety follow-up at the end of treatment 28 days after the last dose, efficacy follow-up every eight weeks, and survival follow-up every three months.

Participants will need to understand the requirements and risks of the trial, sign an informed consent form, accept the dosing regimen required by the trial protocol, and follow the investigator's guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, gender unlimited.
2. Patients with histologically confirmed locally advanced or metastatic solid tumors who have failed standard therapy, are intolerant to standard therapy, or have no standard therapy.

   A. For patients with Non Small Cell Lung Cancer(NSCLC), previous first-line treatment has failed (including chemotherapy or immunotherapy or targeted therapy).

   B. For patients with colorectal cancer, at least previously experienced a systemic treatment regimen (patients with colorectal cancer and high microsatellite instability must have received at least programmed death 1(PD-1) or programmed cell death-Ligand 1(PD-L1) therapy if clinically applicable).

   C. Patients with solid tumors other than NSCLC or colorectal cancer should have received at least systemic therapy and treatment failure.
3. Patients with stage I b are required to have at least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST1.1). Tumor lesions that have previously received radiotherapy or other local treatment are considered measurable lesions only if disease progression at the treatment site is clearly documented after completion of treatment.
4. The ECOG score is 0-1, and there is no decline in physical agility in the two weeks before the first medication.
5. Expected survival is at least 12 weeks.
6. For patients with KRAS G12C mutation, previously confirmed genomic KRAS GI2C mutation results in tumor tissue specimens and hematological specimens were acceptable.
7. Good organ and bone marrow function, provided no blood transfusion has been received within 14 days prior to the screening period, and these results should be completed within 7 days prior to initiation of study therapy:

   1. Bone marrow function should be satisfied: Absolute Neutrophil Count (ANC)≥1.5×10^9/L; Platelet count (PLT)≥100×10^9/L: hemoglobin (Hb)≥9g/dL.
   2. Renal function: serum creatinine (Cr)≤1.5 times the upper limit of normal or creatinine clearance ≥50ml/min as calculated using the Cockcroft-Gault formula.
   3. Liver function: Total bilirubin (TBIL)≤1.5×ULN(TBIL≤2.0×ULN for subjects with documented Gilbert syndrome or TBIL≤3.0×ULN for subjects with indirect bilirubin levels indicating the source of extrahepatic elevation); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×ULN(ALT and AST≤5×ULN if liver metastasis occurs).
   4. Coagulation function: prothrombin time (PT) or partial thromboplastin time (PTT)≤1.5× upper limit of normal (ULN), or international normalized ratio (INR)≤1.5 or within the target range (if prophylactic anticoagulant therapy is performed).
   5. Thyroid function: Thyroid function tests are normal or abnormally asymptomatic and do not require treatment.
8. The elution period of macromolecular drugs and intravenous chemotherapy drugs is ≥4 weeks, and the elution period of oral fluorouracil and small-molecule targeted drugs is ≥2 weeks.
9. For fertile men and women, it is necessary to be willing to use an appropriate contraceptive method 30 days before the first study drug administration and 6 months after the last study drug administration.
10. Did not participate in clinical trial as a subject within 1 month before participating in this trial.
11. Remission to baseline severity or national cancer institute common terminology criteria for adverse events(NCI CTCAE) version 5.0≤ level 1 of all acute toxic reactions from previous anticancer treatments or surgical procedures (except for alopecia or other toxicities deemed by the investigator to be of no safety risk to the patient).
12. Willing to sign informed consent after comprehensive understanding.

Exclusion Criteria:

1. Advanced patients with a short-term risk of life-threatening complications (patients with visceral crisis).
2. Symptomatic or unstable central nervous system(CNS) metastasis, characterized by clinically symptomatic cerebral edema, spinal cord compression, cancerous meningitis, pia meningeal disease, and/or progressive growth. Stable is defined as: 1) seizure-free status continued for >12 weeks with or without antiepileptic drugs; 2) glucocorticoids is not required; 3) Continuously multiple consecutive imaging examinations (scan interval of at least 8 weeks) showed a stable state.
3. Known impairment of gastrointestinal (GI) function or Gl diseases that may significantly affect the absorption or metabolism of oral drugs.
4. Patients who had major surgery (or planned major surgery during the study period), chemotherapy, radiation therapy, any investigational drug, or other anticancer therapy within 4 weeks prior to study entry.
5. Known or suspected allergic symptoms to any component of BEBT-607 tablets.
6. The patient received the following treatments in the 7 days prior to study beginning and plans to use the following drugs throughout the regimen: drugs known to be potent inhibitors/inducers of cytochrome P450 3A4(CYP3A4), cytochrome P450 2C8(CYP2C8), and cytochrome P450 2D6(CYP2D6); Drugs known to significantly lengthen the QT interval.
7. At rest, QT interval (QTc)>470msec(female) or >450msec(male) of Fridericia's mean correction from 3 electrocardiogram (ECG) tests (only retest and take 3 mean corrections if the first ECG indicates QTc>470msec(female) or >450msec(male)); A history of long QT syndrome or a proven long QT synthesis Family history: Clinically significant history of ventricular arrhythmias, or current use of antiarrhythmic drugs or implantation of a defibrillation device for the treatment of ventricular arrhythmias.
8. Uncontrolled electrolyte disturbances may affect the effect of QTc protractive drugs (e.g., hypocalcaemia <1.0mmol/L, hypokalemia < lower limit of normal).
9. Prior combination of severe/unstable angina pectoris, persistent arrhythmia of NCI CTCAE version 5.0≥level 2, atrial fibrillation of any level, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism), myocardial infarction, or coronary/peripheral artery bypass graft within 6 months.
10. Patients with stroke or other severe cerebrovascular disease in the 12 months prior to enrollment.
11. Uncontrolled active severe infections and clinically significant active infections including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related diseases. Active hepatitis B is defined as positive for Hepatitis B surface antigen (HBsAg) and/or Hepatitis Be antigen (HBeAg) with HBV-DNA≥2000IU/ml(equivalent to 10^4 copies /ml); Active hepatitis C is defined as HCV RNA above the upper limit of detection.
12. There is a third space effusion that cannot be controlled by drainage or other methods (such as excessive pleural fluid and ascites).
13. In the investigator's judgment, there are accompanying diseases of seriously patient's safety endangered or patients completing the study affected (such as uncontrolled hypertension, uncontrolled diabetes, severe autoimmune disease, uncontrolled interstitial pneumonia, and thyroid disease).
14. Other severe acute or chronic medical or psychiatric conditions or abnormalities in laboratory tests that may increase the risk of participation in the study or increase the risks associated with the administration of study drugs, or interfere with the study results, and other conditions in which the investigator considers the patient to be unsuitable for participation in the study.
15. Pregnant or lactating women. Defined as women in a state from conception to termination of pregnancy, identified by laboratory human chorionic gonadotropin (hCG) test within 7 days before the start of the study.
16. Recent or active suicidal ideation or behavior.
17. For patients with other malignancies or a history of other malignancies, except for basal cell or squamous cell carcinoma of the skin, papillary carcinoma of the thyroid gland, carcinoma in situ of the cervix and ductal carcinoma in situ of the breast, which has been effectively controlled in the past, is non-invasive and has not recurred or metastasized for 5 years.
18. Difficulty swallowing, or suffering from malabsorption syndrome, or other diseases that are unable to absorb drugs through the intestine or conditions that affect the absorption of BEBT-607.
19. Known active tuberculosis.
20. Patients with Gilbert syndrome or other diseases that may result in an increased susceptibility to abnormal liver function tests during the study period.
21. Other situations judged by the investigator to be ineligible for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
MTD | Phase Ⅰa:Day 2 after the single dose phase, day 1, day 15, and day 28 of the first cycle of the continuous dose phase，assessed up to 4 weeks.
  Maximum tolerated dose
DLT | Phase Ⅰa:Day 2 after the single dose phase, day 1, day 15, and day 28 of the first cycle of the continuous dose phase，assessed up to 4 weeks.
  Dose-limiting toxicity
RDE | Phase Ⅰa:Day 2 after the single dose phase, day 1, day 15, and day 28 of the first cycle of the continuous dose phase，assessed up to 4 weeks.
  Expand the recommended dose
AE | Phase Ⅰa:From the first administration of the study drug to 28 days after the last administration of the study drug.
  Adverse event
ORR | Phase Ⅰb:Every 8 weeks，assessed up to 20 months.
  Objective response rate
PR2D | Phase Ⅰb:Every 8 weeks，assessed up to 20 months.
  Recommended Phase II Dose

SECONDARY OUTCOMES:
PFS | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival
ORR | Phase Ⅰa:Every 4 weeks，assessed up to 4 weeks.
  Objective response rate
DOR | Phase Ⅰa:Every 4 weeks，PhaseⅠb:Every 8 weeks，assessed up to 24 months.
  Duration of response
DCR | Phase Ⅰa:Every 4 weeks，PhaseⅠb:Every 8 weeks，assessed up to 24 months.
  Disease control rate
AE | Phase Ⅰb:From the first administration of the study drug to 28 days after the last administration of the study drug.
  Adverse event
AUC0-t | Phase Ⅰa:Day 1 and Day 28 of cycle 1 before administration and within 48 hours after administration (each cycle is 28 days).Phase Ⅰb:Day 1 and Day 28 of cycle 1 before administration and within 24 hours after administration (each cycle is 28 days).
  Area under the plasma concentration time curve from 0 hour to last time of quantifiable concentration after administration
Cmax | Phase Ⅰa:Day 1 and Day 28 of cycle 1 before administration and within 48 hours after administration (each cycle is 28 days).Phase Ⅰb:Day 1 and Day 28 of cycle 1 before administration and within 24 hours after administration (each cycle is 28 days).
  Peak Plasma Concentration
Tmax | Phase Ⅰa:Day 1 and Day 28 of cycle 1 before administration and within 48 hours after administration (each cycle is 28 days).Phase Ⅰb:Day 1 and Day 28 of cycle 1 before administration and within 24 hours after administration (each cycle is 28 days).
  Time of peak Plasma Concentration
Vss | Day 1 and Day 28 of cycle 1 before administration and within 48 hours after administration,Day 15 and Day 27 of cycle 1 before administration (each cycle is 28 days).
  Apparent volume of distribution
t1/2 | Phase Ⅰa:Day 1 and Day 28 of cycle 1 before administration and within 48 hours after administration (each cycle is 28 days).Phase Ⅰb:Day 1 and Day 28 of cycle 1 before administration and within 24 hours after administration (each cycle is 28 days).
  Half-life of plasma drug concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Heli Liu, Ph.D, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China